CLINICAL TRIAL: NCT06617533
Title: Evaluation of the Primary Care First Model
Acronym: PCF
Status: Active, not recruiting | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MPR50886
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: All Conditions
Keywords: Primary Care First; PCF; primary care delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: PCF practices: This is the intervention group, and includes the practices that were selected and agreed to participate in the PCF model.
  Interventions: Other: PCF model
- No Intervention: Comparison practices: Comparison practices are the control group. This group includes practices not participating in the model that were matched to the PCF practices and whose outcomes will be compared to those of the PCF practices.

INTERVENTIONS:
Other: PCF model — PCF practices practices receive (1) a per-beneficiary-per-month prospective payment that depends on the average health of their attributed Medicare beneficiaries; (2) a Flat Visit Fee for primary care visits, subject to a geographic adjustment factor, and (3) a Performance-based Adjustment (PBA). The PBAs depend on practices' performance on several quality measures in addition to their performance in reducing beneficiaries' use of inpatient care or total cost of care, relative to national and regional benchmarks. Practices must meet a limited set of care delivery requirements and can use the PCF Model's flexible use of payments to invest in strategies that best suit their practices' unique patient population and resources. In return, practices take on limited financial risk in exchange for performance-based payments that reward participants that meet certain performance and quality benchmarks for selected outcomes.
  Groups: Experimental: PCF practices

SUMMARY:
The Primary Care First (PCF) Model, sponsored by the Center for Medicare & Medicaid Innovation (Innovation Center) of the Centers for Medicare & Medicaid Services (CMS), is a multipayer advanced primary care model that aims to strengthen primary care by transforming how primary care practices deliver care. The PCF evaluation will assess how the PCF Model was implemented; how practices transformed care; and the effects on health care cost, service use, quality of care, and the experiences of patients, primary care practitioners, and staff. The evaluation will also identify facilitators and barriers to implementation and improved outcomes.

DETAILED DESCRIPTION:
The Innovation Center launched the PCF Model in 2021. The PCF Model will test whether financial risk and performance-based payments for outcomes, including the acute hospitalization rate, will (1) reduce total Medicare fee-for-service (FFS) expenditures, (2) reduce use of health care services, and (3) preserve or enhance quality of care. The PCF Model will provide payments to participating practices through (i) a per beneficiary per month (PBPM) prospective payment and (2) a Flat Visit Fee, subject to a geographic adjustment factor. PCF practices may further be eligible for a quarterly Performance-based Adjustment (PBA) based on meeting certain performance and quality benchmarks.

The PCF Model builds on principles and experiences from past Innovation Center initiatives, including the Comprehensive Primary Care Initiative, Multi-Payer Advanced Primary Care Practice (MAPCP) demonstration, and Comprehensive Primary Care Plus (CPC+). CMS enrolled practices in the PCF Model in one of two cohorts. Cohort 1 practices participate from January 1, 2021, through December 31, 2025. Cohort 2 practices participate from January 1, 2022, through December 31, 2026. Cohort 2 includes many practices that participated in CPC+. CMS defines a primary care practice under the PCF Model as one or more primary care providers (physician, nurse practitioner, physician's assistant, or clinical nurse specialist) working within the same physical office location or practice site.

The primary goal of the evaluation is to determine whether the PCF Model preserves or enhances quality of care for Medicare FFS beneficiaries and lower expenditures for CMS. The general study design will compare beneficiaries in PCF practices with beneficiaries that receive care at matched comparison practices that aren't participating in PCF but are located in PCF regions. The study will rely on three types of data sources: (1) Medicare FFS claims and enrollment data, (2) payment data for the PCF Model and other CMS programs, and (3) area-level data sets with information on beneficiary and practice characteristics.. Using these data sources, investigators also plan to evaluate the impact of the model on health care service use and a set of secondary outcomes.

ELIGIBILITY:
Practice Inclusion Criteria:

* Are ready to deliver advanced primary care (as measured by questions on the PCF application) when the model launches.
* Located in 1 of 26 PCF regions
* Have at least 125 attributed Medicare FFS beneficiaries
* Have primary care services comprise at least 50 percent of billing, based on revenue, at model launch.
* Start the model using 2015 certified electronic health record technology, enabling exchange of health information with other providers and systems and connection to regional health information exchange.

Beneficiary Inclusion Criteria:

* Be enrolled in both Medicare Parts A and B
* Have Medicare as their primary payer.

Beneficiary Exclusion Criteria:

* Have end stage renal disease
* Currently enrolled in hospice care
* Covered under a Medicare Advantage or other Medicare health plan
* Currently long-term institutionalized
* Currently incarcerated

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of an intervention group comprised of Medicare fee-for-service beneficiaries assigned to PCF practices and a comparison group comprised of Medicare fee-for-service beneficiaries assigned to matched comparison practices.
Sampling Method: Non-Probability Sample
Enrollment: 25000000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute hospitalization rate | 5 years
  Measured per 1,000 beneficiaries per year. Given the model payment structure rewards practices for decreasing hospitalizations, we hypothesize acute hospitalizations are the primary mechanism for reduced expenditures.
Total Medicare Parts A and B expenditures | 5 years
  Measured in dollars per beneficiary per month. Impacts on expenditures are central to CMS's decisions to expand an Innovation Center model and used to determine model PBA payments for practices.

SECONDARY OUTCOMES:
Medical admissions | 5 years
  Measured per 1,000 beneficiaries per year. Evaluations of similar primary care models (such as Comprehensive Primary Care Plus) found participating practices reduced medical admissions. We may expect to see impacts on this before impacts are evident on the broader acute hospitalization measure, which includes surgical admissions.
Outpatient ED visits | 5 years
  Measured per 1,000 beneficiaries per year. Care delivery activities that seek to reduce acute hospitalizations may reduce ED utilization.
Primary-care-substitutable ED visits | 5 years
  Measured per 1,000 beneficiaries per year. Care delivery activities that seek to reduce acute hospitalizations may reduce ED utilization; effects may be concentrated among primary-care-substitutable ED visits.
Proportion of inpatient discharges at the practice that had a 30-day all-cause unplanned readmission | 5 years
  We may expect to see reductions in hospital readmissions through practices' focus on episodic care management.
Proportion of inpatient discharges at the practice with unplanned 30-day acute care | 5 years
  We may expect to see reductions in unplanned acute care (including ED visits, observation stays, and unplanned readmissions) through practices' focus on episodic care management.
Post-acute care (PAC) expenditures per PAC episode | 5 years
  Fewer acute hospitalizations may result in lower total PAC expenditures if savings in higher-cost institutional care (such as skilled nursing facility stays) offset potential cost increases in lower-cost home health expenditures.
Inpatient expenditures | 5 years
  Measured in dollars per beneficiary per month. Fewer acute hospitalizations may result in lower inpatient expenditures, contributing to lower total Medicare FFS expenditures.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Blue, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica Policy Research, Inc., Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT06617533/Prot_SAP_000.pdf